# **Informed Consent Form**

Phase II, Randomized, Placebo-Controlled, Clinical Trial of Genistein in Reducing the Toxicity and Improving the Efficacy of Intravesical Therapy

NCT Number: NCT01489813

Document IRB Approval Date: 8/07/2018

Version Date: 08/02/2018 IRB Form 09052017

# You Are Being Asked to Be in a Research Study

# What Is a Research Study?

The main purpose of research studies is to gain knowledge. This knowledge may be used to help others. Research studies are not intended to benefit you directly, though some might.

# **Do I Have to Do This?**

No. Being in this study is entirely your choice. If you decide to join this study, you can change your mind later on and withdraw from the research study.

Taking part in a study is separate from medical care. The decision to join or not join the research study will not affect your status as a patient.

# What Is This Document?

This form is an informed consent document. It will describe the study risks, procedures, and any costs to you.

This form is also a HIPAA Authorization document. It will describe how your health information will be used and by whom.

Signing this form indicates you are willing to take part in the study and allow your health information to be used.

# What Should I Do Next?

- 1. Read this form, or have it read to you.
- 2. Make sure the study doctor or study staff explains the study to you.
- 3. Ask questions (e.g., time commitment, unfamiliar words, specific procedures, etc.)
- 4. If there will be medical treatment, know which parts are research and which are standard care.
- 5. Take time to consider this, and talk about it with your family and friends.

#### Study No.: IRB00050273

Emory University and Saint Joseph's Hospital Consent to be a Research Subject / HIPAA Authorization

Document Approved On: 8/7/2018

Version Date: 08/02/2018

IRB Form 09052017

<u>Title</u>: Phase II Randomized Placebo-Controlled Clinical Trial of Genistein in Reducing the Toxicity and Improving the Efficacy of Intravesical Therapy

Sponsor-Investigator: Omer Kucuk, MD

<u>Co-Principal Investigator</u>: Viraj Master, MD PhD

**Study Supporter:** DSM Nutritional Products

#### Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

Before making your decision:

- Please carefully read this form or have it read to you
- Please listen to the study doctor or study staff explain the study to you
- Please ask guestions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form you will not give up any legal rights.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

#### **Purpose**

The purpose of this study is to identify the risks and benefits of a taking genistein supplement, I-Cool®, while receiving intravesical therapy to prevent the recurrence of bladder cancer. Genistein is a chemical found in soy beans.

#### **Procedures**

You will be given a brief questionnaire to fill about demographic information and your urinary symptoms. Before your first intravesical therapy you will be randomly assigned to either receive genistein supplement, I-Cool® tablets or a placebo, an inactive substance. You have a 50:50 chance of being in either group, like the flip of a coin. At each treatment visit you will be asked to bring in your pill diary and fill out a questionnaire about your urinary symptoms (either at the visit or via a phone call). A month after you finish your intravesical therapy you will be asked to return to clinic

Study No.: IRB00050273

Document Approved On: 8/7/2018

where you will have a bladder biopsy to see if the intravesical therapy was effective in stopping cancer from coming back in your bladder. You will be asked to fill out the urinary symptoms questionnaire again as well. Also, the research team will also look at your medical records to get more information about your treatment.

## How will my genistein supplement be provided?

The genistein supplement that you will take will be dispensed by the pharmacy and delivered to the principal investigator or study team member. The principal investigator or health care providers on his/her research team will provide the genistein supplement to you. If you have questions about the genistein supplement, you should ask the study doctors.

## **Risks and Discomforts**

There may be side effects from the study drug that are not known at this time. Your condition may not get better, and it may even get worse, as a result of your being in this study. Using the drug may involve risks that are already known, as well as risks which are currently not known. Problems and side effects may occur that are not currently expected and this includes unusual, unexpected, or previously unreported side effects. You should also understand that your cancer symptoms may not be controlled by the study drug used in this study and may even worsen. Different types of side effects may occur in different people. Therefore, it is important that you report all symptoms and side effects that you experience as soon as they occur, whether or not you think they are caused by the study drug. Since genistein reportedly has anti-inflammatory properties, it is unknown whether genistein may reduce the effectiveness of BCG response by decreasing the inflammation associated with the treatment. You will be informed as soon as possible of any new information about this study drug. Additionally, this study involves answering questionnaires which should not take longer than 5 minutes to complete.

#### **Benefits**

This study is not designed to benefit you directly. Your urinary symptoms may improve while you are in this study but they may not, and they may even get worse. This study is designed to learn more about how genistein supplement affects symptoms from intravesical therapy. The study results may be used to help others in the future.

#### Other Treatment Outside this Study

You do not have to be in this study to be treated. You are free to choose not to take part. The study doctor will discuss these with you. You do not have to be in this study to be treated for you condition.

## **Medical Record**

If you have been an Emory and Saint Joseph's Hospital patient before, then you already have an Emory and Saint Joseph's Hospital medical record. If you have never been an Emory and Saint Joseph's Hospital patient, you do not have one. An Emory and Saint Joseph's Hospital medical record will be made for you if an Emory and Saint Joseph's Hospital provider or facility gives you any services or procedures for this study.

Copies of the consent form/HIPAA authorization that you sign will be put in any Emory and Saint Joseph's Hospital medical record you have now or any time during the study.

Emory and Saint Joseph's Hospital may create study information about you that can help with your care. For example, the results of study tests or procedures. These study results will be put in your

Document Approved On: 8/7/2018

Version Date: 08/02/2018

IRB Form 09052017

Emory and Saint Joseph's Hospital medical record. Anyone who has access to your medical records will be able to have access to all the study information placed there. The confidentiality of the study information in your medical record will be protected by laws like the HIPAA privacy rule. State and federal laws may not protect the research information from disclosure.

The results of some study tests and procedures will be used only for research purposes and will *not* be placed in your medical record. For this study, those items include: the questionnaires filled out at weeks 2, 6, and 10 post-operatively.

Tests and procedures done at non-Emory and Saint Joseph's Hospital places may not become part of your Emory and Saint Joseph's Hospital medical record. Also, if you decide to be in this study, it is up to you to let your other health providers know.

## In Case of Injury

If you get ill or injured from being in the study, Emory and Saint Joseph's Hospital will help you to get medical treatment. Emory and Saint Joseph's Hospital and the sponsor have not, however, set aside any money to pay you or to pay for this medical treatment. The only exception is if it is proven that your injury or illness is directly caused by the negligence of an Emory and Saint Joseph's Hospital or sponsor employee. "Negligence" is the failure to follow a standard duty of care.

If you become ill or injured from being in this study, your insurer will be billed for your treatment costs. If you do not have insurance, or if your insurer does not pay, then you will have to pay these costs.

If you believe you have become ill or injured from this research, you should contact Dr. Omer Kucuk at or Dr. Viraj Master at You should also let any health care provider who treats you know that you are in a research study.

## **Costs**

Emory and Saint Joseph's Hospital will pay for the genistein supplement, I-Cool tablets, or the placebo but does not plan to pay for any other items or services that you may receive if you take part in this study.

Emory and Saint Joseph's Hospital will not pay for your regular medical care. If you have insurance, Emory and Saint Joseph's Hospital will submit claims to your insurance for items and services that the sponsor does not cover. Emory and Saint Joseph's Hospital will send in only those claims for items and services that it reasonably believes your insurance will pay and that the sponsor has not paid.

The actual amount that you have to pay depends on whether or not you have health insurance and whether or not that insurance will pay for any research study costs. Generally, insurance companies will not pay for items and services that are required just for a research study. Some insurance companies will not pay for regular medical treatment or treatment for complications if you are in a study. How much you will have to pay for any co-payments, deductibles or co-insurance depends on your plan. Emory and Saint Joseph's Hospital and the sponsor will not pay for these costs.

It is a good idea to contact your insurance provider and tell them you want to be in this research study. Ask them what they will pay for and what they will not pay for. You can also ask the study

Version Date: 08/02/2018 IRB Form 09052017

team for help in figuring out what you will have to pay.

If you do not have insurance, Emory and Saint Joseph's Hospital will review your case as part of its program for low-income patient care. The standard policies of that program will apply. The program will figure out if you have to pay any costs for taking part in the study and what those costs will be.

## Withdrawal from the Study

You have the right to leave a study at any time without penalty.

For your safety, however, you should consider the study doctor's advice about how to go off the study treatment. If you leave the study before the final planned study visit, the researchers may ask you to have some of the final steps done.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

#### **Authorization to Use and Disclose Protected Health Information**

The privacy of your health information is important to us. We call your health information that identifies you, your "protected health information" or "PHI." To protect your PHI, we will follow federal and state privacy laws, including the Health Insurance Portability and Accountability Act and regulations (HIPAA). We refer to all of these laws as the "Privacy Rules." Here we let you know how we will use and disclose your PHI for the main study and for any optional studies in which you may choose to participate.

#### PHI that Will be Used/Disclosed:

The PHI that we will use or share for the main research study includes:

- Medical information about you including your medical history and present/past medications.
- Results of exams, procedures and tests you have before and during the study.
- Laboratory test results.

#### Purposes for Which Your PHI Will be Used/Disclosed:

We will use and share your PHI for the conduct and oversight of the research study. We will use and share your PHI to provide you with study related treatment and for payment for such treatment. We will also use and share your PHI to conduct normal business operations. We may share your PHI with other people and places that help us conduct or carry out the study, such as laboratories, data management centers, data monitors, contract research organizations, Institutional Review Boards (IRBs) and other study sites. If you leave the study, we may use your PHI to determine your health, vital status or contact information. We will use and disclose your PHI for the administration and payment of any costs relating to subject injury from the study.

### Use and Disclosure of Your Information That is Required by Law:

We will use and disclose your PHI when we are required to do so by law. This includes laws that require us to report child abuse or abuse of elderly or disabled adults. We will also comply with legal requests or orders that require us to disclose your PHI. These include subpoenas or court orders.

Version Date: 08/02/2018

IRB Form 09052017

## Authorization to Use PHI is Required to Participate:

By signing this form, you give us permission to use and share your PHI as described in this document. You do not have to sign this form to authorize the use and disclosure of your PHI. If you do not sign this form, then you may not participate in the research study or receive research-related treatment. You may still receive non-research related treatment.

## People Who will Use/Disclose Your PHI:

The following people and groups will use and disclose your PHI in connection with the research study:

- The Principal Investigator and the research staff will use and disclose your PHI to conduct the study and give you study related treatment.
- Emory and Saint Joseph's Hospital may use and disclose your PHI to get payment for study related treatment and to run normal business operations. c
- The Principal Investigator and research staff will share your PHI with other people and groups to help conduct the study or to provide oversight for the study.
- Dr. Omer Kucuk is the Sponsor of the study. The Sponsor may use and disclose your PHI to make sure the research is done correctly and to collect and analyze the results of the research. The Sponsor may disclose your PHI to other people and groups like study monitors to help conduct the study or to provide oversight for the study.
- The research team and the Sponsor may use and disclose your PHI, including disclosure to insurance carriers to administer payment for subject injury.
- The following people and groups will use your PHI to make sure the research is done correctly and safely:
  - Emory and Saint Joseph's Hospital offices that are part of the Human Research Participant Protection Program and those that are involved in study administration and billing. These include the Emory IRB, the Emory Research and Compliance Offices, and the Emory Office for Clinical Research.
  - Government agencies that regulate the research including: Food and Drug Administration
  - Public health agencies.
  - Research monitors and reviewer.
  - Accreditation agencies.
- Sometimes a Principal Investigator or other researcher moves to a different institution. If this happens, your PHI may be shared with that new institution and their oversight offices. PHI will be shared securely and under a legal agreement to ensure it continues to be used under the terms of this consent and HIPAA authorization.

### **Expiration of Your Authorization**

Your PHI will be used until this research study ends.

## **Revoking Your Authorization**

If you sign this form, at any time later you may revoke (take back) your permission to use your information. If you want to do this, you must write:

Dr. Omer Kucuk

Emory University IRB IRB use only

Study No.: IRB00050273

1365 Clifton Road NE Suite B4301 Atlanta, GA 30322

OR

Dr. Viraj Master The Emory Clinic Department of Urology 1365 Clifton Road, Suite B 1400 Altanta, GA 30322

At that point, the researchers would not collect any more of your PHI. But they may use or disclose the information you already gave them so they can follow the law, protect your safety, or make sure that the study was done properly and the data is correct. If you revoke your authorization you will not be able to stay in the study.

Document Approved On: 8/7/2018

Version Date: 08/02/2018

IRB Form 09052017

## Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them.

To maintain the integrity of this research study, you generally will not have access to your PHI related to this research until the study is complete. When the study ends, and at your request, you generally will have access to your PHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you. If it is necessary for your health care, your health information will be provided to your doctor.

We may remove identifying information from your PHI. Once we do this, the remaining information will not be subject to the Privacy Rules. Information without identifiers may be used or disclosed with other people or organizations for purposes besides this study.

## **Contact Information**

Contact Dr. Omer Kucuk at or Dr. Viraj Master at

- if you have any questions about this study or your part in it,
- if you feel you have had a research-related injury or a bad reaction to the study drug, or
- if you have questions, concerns or complaints about the research

Contact the Emory Institutional Review Board at

- if you have questions about your rights as a research participant.
- if you have questions, concerns or complaints about the research.
- You may also let the IRB know about your experience as a research participant through our Research Participant Survey at <a href="http://www.surveymonkey.com/s/6ZDMW75">http://www.surveymonkey.com/s/6ZDMW75</a>.

**Emory University IRB** IRB use only

Study No.: IRB00050273

Document Approved On: 8/7/2018

# **Consent and Authorization**

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed copy of this form. I agree to take part in the study.

| TO BE FILLED ( Please print your name, sign, and date below consent and authorization form, you will not give the signed form to keep. | if you agree to b | e in the main study. By signing this |
|---|---|---|
| Printed Name of Subject | | |
| Signature of Subject | Date | : am / pm<br>Time (please circle) |
| TO BE FILLED OU | JT BY STUDY TE | EAM ONLY |
| Printed Name of Person Obtaining Consent | | |
| Signature of Person Obtaining Consent | <br>Date | : am / pm<br>Time (please circle) |

Version Date: 08/02/2018

IRB Form 09052017